CLINICAL TRIAL: NCT03441347
Title: Neuralgic Amyotrophy: Central Reorganization and Rehabilitation After Peripheral Dysfunction
Acronym: NA-CONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Princess Beatrix Muscle Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 104752
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Neuralgic Amyotrophy; Neuralgic Amyotrophy, Hereditary; Parsonage Turner Syndrome; Brachial Neuritis
Keywords: Physical therapy; Occupational therapy; Rehabilitation; Motor control
MeSH Terms: conditions — Brachial Plexus Neuritis

STUDY DESIGN:
Intervention Model Description: Patients in the experimental arm start the 17 week experimental intervention right after they enter the study. Patients in the second arm first continue to receive their usual care for 17 weeks, after which they also receive the experimental intervention. Both groups are assessed at baseline and after the initial 17 weeks. The second group is assessed a third time, after they have completed the 17-week experimental treatment program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific rehabilitation program (Experimental): Specific, personalized, multidisciplinary rehabilitation program consisting of physical- and occupational therapy.
  Interventions: Behavioral: Specific rehabilitation program
- Usual Care (Other): Usual care for people with neuralgic amyotrophy, may vary per individual
  Interventions: Behavioral: Specific rehabilitation program; Other: Usual Care

INTERVENTIONS:
Behavioral: Specific rehabilitation program — 17-week specific and personalised rehabilitation program. The program starts with a visit to the Plexus out patient clinic in week 1. During this visit, the patient will be examined by a multidisciplinary team, consisting of a rehabilitation physician, neurologist, physical therapist and occupational therapist, which will form a rehabilitation treatment plan. This treatment plan is implemented through 4 weekly sessions in week 2-5, 2 biweekly sessions in week 6-9 and 2 monthly sessions in week 10-17 . Each treatment session involves one hour of physical- and one hour of occupational therapy.
Other: Usual Care — Participants will receive their usual care for 17 weeks, which may vary for each individual
  Arms: Usual Care

SUMMARY:
This study evaluates the effect of a specific, multidisciplinary and personalized rehabilitation program compared to usual care, on motor control and functional disability in patients with neuralgic amyotrophy.

Half of the participants will start with the 17-week specific rehabilitation program while the other half will first continue their usual care for 17 weeks, after which they will also receive the 17-week specific rehabilitation program.

DETAILED DESCRIPTION:
Neuralgic amyotrophy (NA) is a common (incidence 1:1000) peripheral nervous system disorder caused by acute autoimmune inflammation of the brachial plexus, the nerve bundle going to the shoulder and arm. Many NA patients develop abnormal motor control of the shoulder region (i.e. scapular dyskinesia), which persists even after the peripheral nerve damage has recovered. This suggests that persistent scapular dyskinesia in NA may result from (mal)adaptive changes in the central motor system.

Clinical experience shows that the specific, multidisciplinary and personalized rehabilitation program, focused on cognitive motor control can restore scapular dyskinesia in NA patients. This indicates that impairments in the central motor system likely play a role in persistent scapular dyskinesia and that specific rehabilitation may restore any alterations in central motor control.

We hypothesize that the specific rehabilitation program, focused on cognitive motor control is more effective in improving functional disability than usual care and that it can reverse maladaptive changes in central motor control.

ELIGIBILITY:
Inclusion Criteria:

* (Suspected) diagnosis of neuralgic amyotrophy
* In subacute or chronic phase of neuralgic amyotrophy (>2 months after attack onset)
* Right-handed
* Neuralgic amyotrophy predominantly present in right upper extremity
* Presence of scapular dyskinesia

Exclusion Criteria:

* Patients in the acute phase of NA (characterized by severe pain and inflammation of the brachial plexus)
* (Prior) NA attacks of the lumbosacral plexus or the left upper extremity
* Sever comorbidity
* Any (bio)mechanical constraints of the shoulder girdle
* Any other central nervous system, neurological, or neuromuscular disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

PRIMARY OUTCOMES:
Change in Shoulder Rating Questionnaire (SRQ) score from baseline | Baseline (0 weeks) and post-intervention (17 weeks)
  Change in functional (dis)ability of the shoulder, arm and hand measured with the SRQ
Change in brain activity related to central motor control from baseline | Baseline (0 weeks) and post-intervention (17 weeks)
  Change in the magnitudes of mean functional Magnetic Resonance Imaging signal (Blood-oxygen-level dependent (BOLD) activity) related to motor imagery of the affected arm, quantifying changes in central motor control

SECONDARY OUTCOMES:
Change in performance on motor imagery tasks assessing motor control | Baseline (0 weeks), post-intervention (17 weeks)
  Change in performance on motor imagery tasks. Performance is evaluated by means of reaction times and error rates.
Change in Disability of Shoulder, Arm and Hand (DASH) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in functional (dis)ability of the shoulder, arm and hand measured with the DASH
Change in Checklist individual strength - subscale fatigue (CIS-fatigue) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in experienced fatigue
Change in McGill Pain Questionnaire (MPQ) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in nature, intensity, location, course, and effect on daily life of experienced pain
Change in self-efficacy for performing energy conservation strategies assessment (SEPECSA) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in patient's perceived ability to apply energy conservation strategies to their daily life
Change in Utrecht scale for evaluation of rehabilitation-participation (USER-P) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in patient's participation
Change in Pain self efficacy questionnaire (PSEQ) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in confidence people with ongoing pain have in performing activities while in pain.
Change in Patient activation measure (PAM) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in knowledge, skills and confidence in managing one's own health and/or disease
Change in Short-form 36 (SF-36) score from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in experienced health and health related quality of life
Change in serratus anterior muscle strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted with the serratus anterior muscle from baseline, measured when reaching with extended arm and flexed arm
Change in shoulder endorotation strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted while endorotating the shoulder
Change in shoulder exorotation strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted while exorotating the shoulder
Change in key grip strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted while performing a key grip
Change in pinch grip strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted while performing a pinch grip
Change in hand grip strength from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Change in maximal force exerted while performing a hand grip
Change in reachable workspace from baseline | Baseline (0 weeks), post-intervention (17 weeks)
  Reachable workspace is an objective measure of upper extremity impairment. Reachable workspace is quantified by the relative surface area representing the portion of the unit hemisphere that is covered by the hand movements made during a standardized movement protocol which covers cardinal movements of the shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Groothuis, PhD, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

REFERENCES:
- [Background] Ijspeert J, Janssen RM, Murgia A, Pisters MF, Cup EH, Groothuis JT, van Alfen N. Efficacy of a combined physical and occupational therapy intervention in patients with subacute neuralgic amyotrophy: a pilot study. NeuroRehabilitation. 2013;33(4):657-65. doi: 10.3233/NRE-130993. PMID 24004606
- [Derived] Janssen RMJ, Lustenhouwer R, Cup EHC, van Alfen N, Ijspeert J, Helmich RC, Cameron IGM, Geurts ACH, van Engelen BGM, Graff MJL, Groothuis JT. Effectiveness of an outpatient rehabilitation programme in patients with neuralgic amyotrophy and scapular dyskinesia: a randomised controlled trial. J Neurol Neurosurg Psychiatry. 2023 Jun;94(6):474-481. doi: 10.1136/jnnp-2022-330296. Epub 2023 Jan 25. PMID 36697215
- [Derived] Lustenhouwer R, Cameron IGM, van Alfen N, Toni I, Geurts ACH, van Engelen BGM, Groothuis JT, Helmich RC. Cerebral Adaptation Associated with Peripheral Nerve Recovery in Neuralgic Amyotrophy: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2023 Jan;37(1):3-15. doi: 10.1177/15459683221145149. Epub 2022 Dec 27. PMID 36575812
- [Derived] Lustenhouwer R, van Alfen N, Cameron IGM, Toni I, Geurts ACH, Helmich RC, van Engelen BGM, Groothuis JT. NA-CONTROL: a study protocol for a randomised controlled trial to compare specific outpatient rehabilitation that targets cerebral mechanisms through relearning motor control and uses self-management strategies to improve functional capability of the upper extremity, to usual care in patients with neuralgic amyotrophy. Trials. 2019 Aug 7;20(1):482. doi: 10.1186/s13063-019-3556-4. PMID 31391076